CLINICAL TRIAL: NCT07387991
Title: Clinical Trial to Evaluate the Ability of Multi-Strain Postbiotic to Impact Inflammation, Immune Components, Gastrointestinal Symptoms, Recovery, Anxiety, and Intestinal Permeability
Brief Title: Evaluating the Ability of a Multi-Strain Postbiotic to Impact Inflammation, Immune Components, Gastrointestinal Symptoms, Recovery, Anxiety, and Intestinal Permeability
Acronym: BIO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lindenwood University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB-26-17
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Inflammation; Gastrointestinal Symptoms
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: This study uses a randomized, double-blind, placebo-controlled, parallel-group design. Eligible participants will be randomly assigned to receive either a multi-strain postbiotic supplement or a matched placebo for 28 consecutive days. Randomization will be stratified by sex and age. Participants will remain in their assigned intervention group for the duration of the study.
  At the end of the supplementation period, all participants will complete a standardized 45-minute treadmill exercise bout at 72 to 78% of predicted maximum heart rate to induce a controlled physiological stress. Biological, gastrointestinal, and psychological responses will be assessed before and after the exercise bout to compare responses between the postbiotic and placebo groups.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postbiotic (Experimental): Participants assigned to the postbiotic group will consume a multi-strain postbiotic supplement daily for 28 consecutive days prior to completing a standardized treadmill exercise bout. The supplement will be provided in capsule form and consumed once daily with approximately eight ounces of water.
  Interventions: Dietary Supplement: Multi-Strain Postbiotic
- Placebo (Placebo Comparator): Participants assigned to the placebo group will consume a placebo consisting of microcrystalline cellulose in capsule form daily for 28 consecutive days prior to completing a standardized treadmill exercise bout. The placebo capsules will be identical in size, color, and appearance to the postbiotic capsules and will be consumed once daily with approximately eight ounces of water.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Multi-Strain Postbiotic — Participants will ingest a multi-strain postbiotic supplement once daily for 28 days. Each dose will be consumed with approximately eight ounces of water at the same time each day. If a dose is missed, participants will be instructed to take the missed dose the following day by splitting the dose into one capsule in the morning and one capsule in the evening.
  Arms: Postbiotic
Dietary Supplement: Placebo — Participants will ingest a placebo consisting of microcrystalline cellulose in capsule form once daily for 28 days. The placebo capsules will be identical in size, color, and appearance to the active supplement and will be consumed with approximately eight ounces of water at the same time each day. If a dose is missed, participants will be instructed to take the missed dose the following day by splitting the dose into one capsule in the morning and one capsule in the evening.
  Arms: Placebo

SUMMARY:
This study will evaluate the effects of a multi-strain postbiotic supplement on markers of inflammation, immune function, gastrointestinal symptoms, psychological well-being, and intestinal permeability in healthy adults. The primary objective is to determine whether four weeks of postbiotic supplementation alters physiological and perceptual responses to a standardized bout of moderate-to-high intensity exercise compared with placebo.

Approximately 50 healthy men and women aged 18 to 55 years will be enrolled in a randomized, double-blind, placebo-controlled, parallel-group clinical trial. Participants will be randomly assigned to receive either a multi-strain postbiotic supplement or a matched placebo for 28 days.

At the end of the supplementation period, participants will complete a 45-minute treadmill exercise bout at 75% of their individually determined maximum heart rate. Blood samples will be collected to assess biomarkers of inflammation, immune activity, and recovery. Gastrointestinal symptoms, intestinal permeability, anxiety, and perceived recovery will be evaluated using validated questionnaires.

This study is designed to determine whether postbiotic supplementation modulates physiological stress responses and subjective well-being following prolonged exercise in healthy adults.

DETAILED DESCRIPTION:
This study is designed to evaluate the effects of a multi-strain postbiotic supplement on physiological, gastrointestinal, and psychological responses to a standardized bout of aerobic exercise in healthy adults. Prolonged moderate-to-high intensity exercise is known to acutely increase inflammatory activity, alter immune function, disrupt gastrointestinal integrity, and influence perceptions of recovery and anxiety. Nutritional interventions that can modulate these responses may be beneficial for supporting health and resilience in physically active populations. Postbiotics, which consist of non-viable microbial cells and their metabolic byproducts, have been proposed to influence immune and gastrointestinal function while avoiding some of the stability and safety concerns associated with live probiotics.

Approximately 50 healthy men and women aged 18 to 55 years will be recruited to participate in a randomized, double-blind, placebo-controlled, parallel-group clinical trial. Eligible participants will be randomly assigned to receive either a multi-strain postbiotic supplement or a matched placebo for 28 consecutive days. Both participants and investigators will remain blinded to treatment assignment for the duration of the study.

Participants will be instructed to maintain their habitual diet, physical activity, and lifestyle behaviors throughout the supplementation period and to avoid the use of additional probiotic, prebiotic, or immune-modulating supplements. Compliance with supplementation will be monitored by self-report and capsule counts.

At the end of the 28-day supplementation period, participants will complete a standardized 45-minute treadmill exercise bout performed at 75% of their individually determined maximum heart rate. This exercise protocol is designed to induce a controlled physiological stress that elicits measurable inflammatory, immune, and gastrointestinal responses.

Blood samples will be collected to assess biomarkers related to inflammation, immune function, and recovery. Gastrointestinal symptoms, intestinal permeability, anxiety, and perceived recovery will be assessed using validated questionnaires administered before and after the exercise challenge.

Safety will be monitored throughout the study through the collection of self-reported adverse events and investigator assessment.

This study will determine whether supplementation with a multi-strain postbiotic alters physiological and perceptual responses to prolonged aerobic exercise compared with placebo in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

Healthy males and females aged 18 to 55 years of age. Individual indicates they are physically active defined as: 30 minutes of moderate intensity activity 4 days per week in the past 3 months.

Subject has the ability to exercise on a treadmill without issue or concern. Body Mass Index (BMI) 18.0-32.0 kg/m2 (normal weight to obesity weight). The average BMI of the entire cohort will be <30.0 kg/m2.

Subject is in good health and appropriate for exercise as determined by physical examination and medical history.

Subject can exercise on a treadmill without issue or concern. Subject is a non-smoker. Subject agrees to not use any new vitamin, mineral, or dietary supplements 24 hours prior to the exercise test visits.

Subject is willing and able to comply with the protocol including: attending the study scheduled appointments, of which two of the study visits may take up to four hours of completion.

Subject agrees to refrain from exercise for the 24 hours prior to any test visits.

Subject agrees to refrain from alcohol use for at least 24 hours before every study visit.

Subject is able to understand and sign the informed consent to participate in the study.

Exclusion Criteria:

Individuals who are determined to have liver, renal, cardiovascular, or other metabolic disease.

Use of any dietary supplements, prescription mediation (particularly antibiotics and/or anti-inflammatories), or probiotics within the past 2 months which may confound the study or its endpoints.

Alcohol consumption (>2 standard alcoholic drinks/day or >10 drinks/week) or drug abuse/dependence.

Smokers (defined as greater than 2 cigarettes per day for past 90 days). Clinically significant abnormal laboratory results at screening. Allergy or sensitivity to study supplement ingredients. Individuals who are cognitively impaired and/or who are unable to give informed consent.

Individuals with diabetes, asthma, rheumatoid arthritis, colitis, IBS/IBD, gout, or fibromyalgia.

Any other condition which in the PI's opinion may adversely affect the subject's ability to complete the study, its measurement or poses significant risk to the subject.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Interleukin-6 (IL-6) | Serum IL-6 concentrations will be measured using multiplex bead-based assays to assess the inflammatory response to a standardized 45-minute treadmill exercise bout following 28 days of supplementation.
  Baseline, pre-exercise, immediately post-exercise, 1-hour post-exercise, 3-hours post-exercise, and 24-hours post-exercise after 28 days of supplementation
Tumor Necrosis Factor-α (TNF-α) | Serum TNF-α concentrations will be measured using multiplex bead-based assays to assess exercise-induced inflammatory responses following supplementation.
  Baseline, pre-exercise, immediately post-exercise, 1-hour post-exercise, 3-hours post-exercise, and 24-hours post-exercise after 28 days of supplementation
Interleukin-10 (IL-10) | Serum IL-10 concentrations will be measured to assess anti-inflammatory and immune regulatory responses to exercise following supplementation.
  Baseline, pre-exercise, immediately post-exercise, 1-hour post-exercise, 3-hours post-exercise, and 24-hours post-exercise after 28 days of supplementation
Perceived Recovery Scale (PRS) | Baseline, pre-exercise, immediately post-exercise, 1-hour post-exercise, 3-hours post-exercise, and 24-hours post-exercise
  Subjective recovery will be assessed using the Perceived Recovery Scale (PRS), a 0-10 scale reflecting perceived readiness and recovery status.

CONTACTS AND LOCATIONS:
Overall Officials: Chad M Kerksick, PhD, Principal Investigator — Lindenwood University
Locations (1):
- Exercise and Performance Nutrition Laboratory, Saint Charles, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Data contain sensitive longitudinal biological and symptom information that cannot be reliably de-identified without compromising participant privacy.